CLINICAL TRIAL: NCT06230874
Title: Effectiveness of Mindfulness Protocols Among Occupational Therapy Students
Brief Title: Effectiveness of Mindfulness Protocols Among OT Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeanne Sowers (Other)
Responsible Party: Sponsor-Investigator, Jeanne Sowers, Program Director, Huntington University
Organization: Huntington University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HuntingtonU
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Mindfulness Protocols
Keywords: Mindfulness; Stress; Engagement; Student; Occupation

STUDY DESIGN:
Intervention Model Description: Study participants will be randomly assigned to one of two groups in parallel for the duration of the study.
Who Masked: Participant, Investigator
Masking Description: Individual participants will only have knowledge of their own intervention protocol. The investigators will be blinded to the randomization process and will not have knowledge of the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HOME Protocol (Experimental): Will receive the HOME Protocol Intervention
  Interventions: Behavioral: HOME Protocol
- Control Journaling Protocol (Active Comparator): Will receive the Control Journaling Protocol
  Interventions: Behavioral: Control Journaling Protocol

INTERVENTIONS:
Behavioral: HOME Protocol — The HOME Protocol is a newly developed nine-minute mindfulness and engagement protocol designed to decrease stress and to promote re-engagement in meaningful occupations of daily life by applying mindfulness strategies in a specific, timed format. The protocol requires special training for students: a) to recognize times of disengagement in occupations, and b) to learn how to apply specific mindfulness strategies to increase re-engagement in meaningful occupations. Five components of the HOME Protocol include Reflect (1 minute of self-reflection and self-talk), Reset (2 minutes for breathing with stillness/silence and body check), Reach (3 minutes for stretching and progressive muscular relaxation), Renew (2 minutes for breathing with meditation/gratitude), and Re-engage (1 minute for self-reflection and self-talk).
  Arms: HOME Protocol
Behavioral: Control Journaling Protocol — The control journaling protocol is a nine-minute mindfulness and engagement protocol designed to decrease stress and to promote re-engagement in meaningful occupations of daily life by applying mindfulness self-talk and journaling strategies in a specific, timed format. The protocol requires special training for students: a) to recognize times of disengagement in occupations, and b) to learn how to apply specific mindfulness strategies to increase re-engagement in meaningful occupations. Three components of the control journaling protocol include Reflect (1 minute of self-reflection and self-talk), Write (journaling), and Re-engage (1 minute for self-reflection and self-talk).
  Arms: Control Journaling Protocol

SUMMARY:
The research will study the effectiveness of mindfulness protocols for OT students to decrease stress and re-engage in meaningful occupations after becoming disengaged.

DETAILED DESCRIPTION:
The current study aims to investigate the effectiveness of a mindfulness protocol for OT students to decrease stress and reengage in meaningful occupations after becoming disengaged.

Anticipated benefits for participants include learning mindfulness techniques that may aid in stress reduction and promotion of re-engagement in meaningful occupations, such as schoolwork. Additionally, the results of this study can provide future OT students with information related to the effectiveness of mindfulness and re-engagement protocol.

Procedures:

Recruitment:

The research team will attempt to recruit at least 50 participants for this study using convenience and snowball sampling methods. An email invitation with a recruitment flyer will be sent to program directors of accredited entry-level graduate OT programs in the continental United States to invite potential participants interested in the study. Snowball sampling methods will also be utilized by sharing the recruitment flyer on OT social media sites, and through email to student representatives of OT associations and to faculty and student contacts. A Formstack link will be provided in the email invitation for interested participants to complete a short survey to determine if they meet the inclusion criteria. Participants must voluntarily sign a consent form on Formstack to participate in the study. Recruitment will begin following IRB committee approval and continue until mid-January 2024.

Enrollment:

Immediately following the recruitment period, voluntary participants that meet the inclusion/exclusion criteria on an interest survey and complete the voluntary consent form via Formstack will be enrolled in the study. Study participants will be given a numerical identifier for the duration of the research study. The investigators will be blinded to participants' names prior to randomizing the sample. The research support team will randomize the sample into one of two groups (experimental and control) utilizing a random number generator. The investigators will not have knowledge of the interventions assigned to individual participants.

Data Collection:

Following randomization, the participants will be emailed with their numerical identifier and information on how to access the pre assessments. Pre assessments will include a demographic survey, the COPE Inventory, and the PSS. Following completion of the pre assessments, participants will be given information on how to access their designated virtual mindfulness training (experimental or control). The experimental group will complete a 1-1.5 hour training in the use of the HOME Protocol, which was developed and pilot tested. The control group will complete an alternate 1-1.5 hour training in mindfulness that focuses on self-talk and journaling strategies. The mindfulness trainings were originally developed in 2020 by Huntington University OTD faculty and students and have been updated by the current researchers for use in this study. Scripts written by the researchers will be used in each training to ensure standardization for future studies. The timeframe for each virtual training will take 1-1.5 hours. Upon completion of the virtual training, participants will utilize their specific mindfulness protocol in accordance with the training received. Each protocol will take nine minutes to complete. The participants will be asked to complete their designated research protocol checklist using a virtual platform at least once a week for four weeks. Participants will record their perceived levels of stress, engagement, difficulty and meaningfulness of the activity, and other feelings before and after each use of their respective protocol checklist via a virtual survey platform. Participants will be sent weekly email reminders to complete their mindfulness protocols and checklists during the 4-week intervention period.

At the end of the four-week intervention period, participants will be emailed information on how to access the post assessments, which include the PSS and the COPE Inventory.

Participants will be incentivized with a random drawing consisting of two $50 gift cards for completing the entirety of the research study. Only the names of participants who complete their respective mindfulness protocol a minimum of once per week for four weeks and complete the 1-1.5 hour virtual training and pre and post assessments will be included for the random incentive drawing that will occur at the end of the intervention and data collection period. Participants that complete the entirety of the study will also be offered the opportunity to receive a 1-1.5 hour virtual training in the alternate mindfulness protocol approximately one month following the completion of the research.

Data analysis and Hypotheses:

Pre and post assessment data of the PSS and COPE Inventory will be analyzed for significant changes from pre assessment to post assessment scores and responses. Data from the experimental and control group protocol checklists will be compiled and analyzed for significant changes during the intervention process.

Following 4 weeks of protocol use, the null hypotheses propose: no statistically significant differences between the experimental and control groups for the Perceived Stress Scale (PSS) and the Coping Orientation to Problems Experienced (COPE) Inventory change scores pre and post intervention. Additionally, to determine the immediate effect of protocol use, the change scores of the protocol checklist Likert scales collected in the first and last minutes during the 9-minute protocol will be examined. Data from week 4 will be used because the participants will be most familiar with their protocol use by this time. The null hypotheses propose: no statistically significant differences between experimental and control groups for the protocol checklist Likert scales stress or engagement change scores in week 4; and no statistically significant differences within groups for reported stress or engagement immediately after the use of the protocol in week 4. The alpha level is set at 0.01.

During the data collection and analysis process, all participants will be assigned a numeric identifier and de-identified data will be kept private on password-protected computers using Excel or a similar platform. A master list of the participants in the experimental and control groups with their corresponding email and numerical identifiers will be printed and kept in a locked box in a secure cabinet on the 3rd floor of the Huntington University OTD Program at 1819 Carew St., Fort Wayne, IN 46805. The master list will be kept private and separate from the numerical data. All electronic data, including data sets from the pre and post assessments, and protocol data, will be stored for a minimum of three years on an OTD program password-protected computer. All printed data will be kept for a minimum of three years in a secure cabinet of the Huntington University OTD Program.

This study presents minimal risks to participants. The greatest risk is emotional distress participants may feel related to self-reflection on stress levels. Additionally, there is a time requirement for virtual completion of the training, protocol checklists, and pre/post assessments.

Researchers have attempted to reduce potential risk by keeping the length of the virtual training to 1-1.5 hours. Additionally, the participants' mindfulness protocols will require only 9 minutes to complete and at a minimum of once a week for four weeks. There is a potential risk for a breach of confidentiality due to the use of virtual training and electronic data collection methods. The researchers have attempted to reduce risk by utilizing numerical identifiers throughout the research process. Subject numbers will be kept on a private confidential master list to ensure anonymity.

ELIGIBILITY:
Inclusion Criteria

* 18 years or older
* Currently in an accredited entry-level graduate OT program in the continental United States
* Must complete pre and post assessments.
* Must complete a one-time 1-1.5-hour virtual mindfulness training.
* Must utilize the mindfulness research protocol for at least once a week for a four-week period.

Exclusion Criteria:

* Under 18 years
* Not enrolled in an accredited entry-level graduate OT program in the continental US.
* Must complete pre and post assessments.
* Must complete a one-time 1-1.5-hour virtual mindfulness training
* Must utilize research protocol at least once a week for a four-week period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | Through study completion, up to two weeks
  The PSS is a questionnaire composed of 10 questions to assess perceptions of stress and the degree to which one perceives life situations as stressful. Literature supports the PSS as a valid and reliable assessment of perceived stress of university students.
Coping Orientation to Problems Experienced (COPE) Inventory | Through study completion, up to two weeks
  The COPE is self-report instrument composed of 60 questions to assess people's stress responses. For this study, we will use the behavioral disengagement and mental disengagement scales to measure the participants' response to stress prior to and following the intervention period.
Protocol Checklist | Week 4 Data
  Each protocol (HOME Protocol and Control Journaling Protocol) has a checklist that is embedded in the protocol measures the student's perceived level of stress, engagement, challenge, and meaning of the activity that they disengage from. Four Likert rating scales (0 representing the lowest score and 10 representing the highest score) are embedded in the first minute and final minute of the protocol to record students' self-assessments pre and post intervention in the following areas: stress, engagement, challenge, and meaning. By the 4th week of the intervention the student participants are most likely to have learned to use their respective protocols; therefore, the study will utilize only week 4 protocol data to determine between group and within group differences of the stress and engagement scale change scores immediately following use of the protocols.

CONTACTS AND LOCATIONS:
Locations (1):
- Huntington University, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerig, L., Henton, P., Butterweck, M., Swider, J., Cameron, L., Marihugh, K., & Close, K. (2023). Stress, Mindfulness and Occupational Engagement: A Pilot Study of the HOME Protocol. Journal of Occupational Therapy Education, 7 (2). https://doi.org/10.26681/jote.2023.070204
- [Background] Carver CS, Scheier MF, Weintraub JK. Assessing coping strategies: a theoretically based approach. J Pers Soc Psychol. 1989 Feb;56(2):267-83. doi: 10.1037//0022-3514.56.2.267. PMID 2926629
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Cohen, S., & Williamson, G. (1988). Perceived stress in a probability sample of the United States. In S. Spacapam & S. Oskamp (Eds.) The Social Psychology of Health (pp. 31-67). Sage Publications.
- [Background] Lee EH. Review of the psychometric evidence of the perceived stress scale. Asian Nurs Res (Korean Soc Nurs Sci). 2012 Dec;6(4):121-7. doi: 10.1016/j.anr.2012.08.004. Epub 2012 Sep 18. PMID 25031113
- [Background] Roberti, J. W., Harrington, L. N., & Storch, E. A. (2006). Further psychometric support for the 10-item version of the Perceived Stress Scale. Journal of College Counseling, 9(2), 135-147. https://doi.org/10.1002/j.2161-1882.2006.tb00100.x